CLINICAL TRIAL: NCT07303894
Title: Randomized, Multi-dose, Placebo-controlled Phase 2 Trial of Oral Isoquercetin to Reduce Thrombin Generation in Ovarian Cancer
Brief Title: A Study of Isoquercetin in People With Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-060
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer; Epithelial Ovarian Cancer; Serous Ovarian Tumor
Keywords: Ovarian Cancer; Epithelial Ovarian Cancer; Serous Ovarian Tumor; Isoquercetin; Memorial Sloan Kettering Cancer Center; 25-060
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — isoquercitrin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Cohort B: Isoquercetin daily (Experimental)
  Interventions: Drug: Isoquercetin
- Cohort C: Isoquercetin twice daily (Experimental)
  Interventions: Drug: Isoquercetin

INTERVENTIONS:
Drug: Isoquercetin — Cohort B and Cohort C will take isoquercetin
  Arms: Cohort B: Isoquercetin daily; Cohort C: Isoquercetin twice daily
Other: Placebo — Placebo
  Arms: Cohort A: Placebo

SUMMARY:
The purpose of this study is to test whether isoquercetin can reduce markers in the blood that may indicate the risk of blood clots in people with ovarian cancer. The effects of isoquercetin will be compared with those of a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histological- or cytological-confirmed ovarian cancer (epithelial, serous, or clear cell) and be receiving first-line chemotherapy (day 1 of isoquercetin should align with day 1 of cycle 1 or 2 of chemotherapy) for neoadjuvant, adjuvant, or advanced settings.
* Minimum age 18 years
* Life expectancy of greater than 6 months.
* ECOG performance status <2
* Participants must have preserved organ and marrow function as defined below:

  * Platelet count > 50,000/mcL
  * Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.5 x institutional upper limit of normal (ULN)
  * Total bilirubin < 3 x ULN without liver metastases and <5 x ULN in presence of liver metastases.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 X ULN without liver metastases and <5 x ULN in the presence of liver metastases.
  * Estimated creatinine clearance (CrCl >30 ml/min)
* The effects of isoquercetin on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior history of documented venous thromboembolic event within the last 2 years (excluding central line associated events whereby patients completed anticoagulation)
* Active bleeding or high risk for bleeding (e.g., known acute gastrointestinal ulcer)
* History of significant hemorrhage (requiring hospitalization or transfusion) outside of a surgical setting within the last 24 months
* Familial bleeding diathesis
* Known diagnosis of disseminated intravascular coagulation (DIC)
* Currently receiving anticoagulant therapy
* Current daily use of aspirin, clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox) (within 10 days) or considered to use regular use of higher doses of non-steroidal anti-inflammatory agents as determined by the treating physician (e.g ibuprofen > 800 mg daily or equivalent)
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known intolerance of (iso)quercetin, niacin or ascorbic acid (including known G6PD deficiency).
* Participants with known brain metastases
* Pregnant women are excluded from this study because isoquercetin is a PDI inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with isoquercetin, breastfeeding should be discontinued if the mother is treated with isoquercetin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Level of PDI-sensitive, platelet-dependent thrombin generation measured as compared to baseline | up to 6 weeks from baseline
  The primary endpoint is the maximal inhibition of PDI-sensitive, platelet-dependent thrombin generation measured at either 3 or 6 weeks (relative to baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zwicker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Beth Israel Deaconess Medical Center (Data Collection Only), Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities ), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org